CLINICAL TRIAL: NCT02712580
Title: Clinical Trial for Therapeutic Effect of Wireless Micro Current Stimulation Under Objectification of Combustion Depth by Laser Doppler Imaging in Children and Adolescents With Deep Dermal Burns and Scald Injuries
Brief Title: Therapeutic Effect of the Wireless Micro Current Stimulation in Pediatric Deep Dermal Burns and Scald Injuries
Acronym: ELSTHER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kinderkrankenhaus auf der Bult (Other)
Responsible Party: Principal Investigator, Mechthild Sinnig, MD, Head of burn center, Principal Investigator, Kinderkrankenhaus auf der Bult
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1234567
Record Dates: First submitted 2016-01-04; First posted 2016-03-18 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Burns
Keywords: pediatric burns; deep dermal wounds; wound healing; ChildPain Measurement; Treatment Outcome Wound Healing/physiology; wireless electric stimulation; wireless current stimulation; wireless technology; children; conservative treatment; deep dermal scalds; humans; deep dermal burns; burns; wound healing process
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- First investigational device (Active Comparator): official name of product: "Wireless microcurrent Stimulation Wetling W 200" n=47 patients The irradiation time is 30 minutes a day, the depth of penetration of the electrons in the skin stimulation is 1.5 uA. The irradiation is accompanied by white light.
  Interventions: Device: First investigational device
- Second investigational device (Active Comparator): official name of product: "Wireless microcurrent Stimulation Wetling W 200" n=47 patients The irradiation time is 30 minutes a day, the depth of penetration of the electrons in the skin stimulation is 1.5 uA. The irradiation is accompanied by red light.
  Interventions: Device: Second investigational device
- ES Wetling W200 with white light (Placebo Comparator): Placebo device - 'ES Wetling W200 Placebo with white light' n=47 patients The placebo-irradiation time is 30 minutes a day. The placebo irradiation is accompanied by white light.
  Interventions: Device: ES Wetling W200 Placebo with white light
- ES Wetling W200 with red light (Placebo Comparator): Placebo device - 'ES Wetling W200 Placebo with red light' n=47 patients The placebo-irradiation time is 30 minutes a day. The placebo irradiation is accompanied by red light.
  Interventions: Device: ES Wetling W200 Placebo with red light

INTERVENTIONS:
Device: First investigational device — The irradiation time is 30 minutes a day, the depth of penetration of the electrons in the skin stimulation is 1.5 uA. The irradiation is accompanied by white light.
  Other Names: Wireless microcurrent Stimulation Wetling W 200
  Arms: First investigational device
Device: Second investigational device — The irradiation time is 30 minutes a day, the depth of penetration of the electrons in the skin stimulation is 1.5 uA. The irradiation is accompanied by red light.
  Other Names: Wireless microcurrent Stimulation Wetling W 200
  Arms: Second investigational device
Device: ES Wetling W200 Placebo with white light — The placebo-irradiation time is 30 minutes a day. The placebo irradiation is accompanied by white light.
  Other Names: non-invasive Electrical Stimulation Lamp
  Arms: ES Wetling W200 with white light
Device: ES Wetling W200 Placebo with red light — The placebo-irradiation time is 30 minutes a day. The placebo irradiation is accompanied by red light.
  Other Names: non-invasive Electrical Stimulation Lamp
  Arms: ES Wetling W200 with red light

SUMMARY:
This study will determine the effect of the wireless micro current stimulation in pediatric deep dermal burns and scald injuries. The clinical trial ist designed as a blinded, placebo-controlled, randomized, prospective, single-center study.

DETAILED DESCRIPTION:
Patients (m / w) aged 0-17 years with scalding and burning injuries will initially receive polyhexanide gel 0.02% in the ordinary course.

After 24-48 hours after the accident the wound depth is measured and documented with laser Doppler imaging (see inclusion criteria).

Then the patient is enclosed into the study.

From day 3 after the accident daily dressing changes are performed with possibly slight analgesic medication (ibuprofen 10 mg / kg ) and if necessary under sedation with midazolam 0.5 mg / kg po. Here, a 30-minute-treatment with the wireless micro current stimulation or the placebo lamp is performed.

For visual support of the process of the colorless wireless microcurrent therapy / colorless placebo therapy the medical device has an additional light source (red and white color). So, in addition, both (the control and the placebo) groups are divided in one group with colorless intervention (white light) and a group with red light. The main aspect is to avoid bias.

The treated wound areas are examined daily during the dressing change by the study doctors and standardized photographed.

The condition of the wound is detected in the wound documentation module of KIS. The end point of the wireless micro current stimulation is an epithelialization of the wound surface under investigation of> 95%. The detection of reepithelisation is performed by the investigators and objectified through a photo-image program.

At the total absence of wound healing on day 16th, the patient receives the standard surgical therapy (skin grafting).

If there is an absence of wound healing with less than 50% epithelisation after 3 weeks of wireless micro current stimulation therapy the patient will also receives the standard surgical treatment (skin graft).

If the wound-epithelialisation at day 24 is greater than 50% but not> 95%, the wireless micro current stimulation will still be continued, but no longer than 4 weeks - until day 30.

ELIGIBILITY:
Inclusion Criteria:

* inpatients (m / w)
* wound area greater than 0.5% and less than / or equal to 3% of the body surface
* IIb ° combustion depth verified by Laser Doppler Imaging
* Burn / scalds not older than 48 hours
* Participation willingness of the patient
* willingness to participate and written informed consent of both parents (or legal guardian) of the patient

Exclusion Criteria:

* known wound healing problems
* child abuse as the cause of the combustion
* different wound dressing treatment prior to transfer to our hospital

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 188 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Epithelialization of the examined wound area of> 95% | up to 30 days
  The primary endpoint of the trial is a epithelialization of the examined wound area of> 95%. The primary endpoint is the time to reach a epithelialization of the wound defect> 95%, measured in days since initial treatment (= initial treatment of the wound). In absence of wound healing after initial treatment and study treatment, the then usual surgical treatment for deep dermal wounds will be performed in patients (skin graft).

SECONDARY OUTCOMES:
Pain measurements | up to 21 days
  The secondary endpoints include the subjective pain. This is detected every 8 hours (starting at 8:00 am) during hospitalization and indicated by a validated, visual analogue pain scale through study completion
Pain killer consumption | up to 21 days
  The painkiller consumption per kg / body weight and day is captured through study completion

CONTACTS AND LOCATIONS:
Overall Officials: Mechthild Sinnig, MD, Principal Investigator — Kinder- und Jugendkrankenhaus AUF DER BULT
Locations (1):
- Pediatric Surgery Kinder- und Jugendkrankenhaus AUF DER BULT, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albertini R, Villaverde AB, Aimbire F, Salgado MA, Bjordal JM, Alves LP, Munin E, Costa MS. Anti-inflammatory effects of low-level laser therapy (LLLT) with two different red wavelengths (660 nm and 684 nm) in carrageenan-induced rat paw edema. J Photochem Photobiol B. 2007 Nov 12;89(1):50-5. doi: 10.1016/j.jphotobiol.2007.08.005. Epub 2007 Sep 6. PMID 17920925
- [Background] Cramp AF, Noble JG, Lowe AS, Walsh DM. Transcutaneous electrical nerve stimulation (TENS): the effect of electrode placement upon cutaneous blood flow and skin temperature. Acupunct Electrother Res. 2001;26(1-2):25-37. doi: 10.3727/036012901816356036. PMID 11394491
- [Background] Cho MR, Thatte HS, Lee RC, Golan DE. Integrin-dependent human macrophage migration induced by oscillatory electrical stimulation. Ann Biomed Eng. 2000 Mar;28(3):234-43. doi: 10.1114/1.263. PMID 10784088
- [Background] Goldman RJ, Brewley BI, Golden MA. Electrotherapy reoxygenates inframalleolar ischemic wounds on diabetic patients: a case series. Adv Skin Wound Care. 2002 May-Jun;15(3):112-20. doi: 10.1097/00129334-200205000-00006. PMID 12055444
- [Background] Fiorio FB, Silveira L Jr, Munin E, de Lima CJ, Fernandes KP, Mesquita-Ferrari RA, de Carvalho Pde T, Lopes-Martins RA, Aimbire F, de Carvalho RA. Effect of incoherent LED radiation on third-degree burning wounds in rats. J Cosmet Laser Ther. 2011 Dec;13(6):315-22. doi: 10.3109/14764172.2011.630082. PMID 21981305
- [Background] Herberger K, Kornek T, Debus ES, Diener H, Augustin M. Electrotherapy of chronic wounds: evidence of clinical effectiveness and benefit. Wound Manage 2011;2:86 - 93.
- [Background] Kaada B, Olsen E, Eielsen O. In search of mediators of skin vasodilation induced by transcutaneous nerve stimulation: III. Increase in plasma VIP in normal subjects and in Raynaud's disease. Gen Pharmacol. 1984;15(2):107-13. doi: 10.1016/0306-3623(84)90091-0. PMID 6714637
- [Background] Kamolz, Herndon, Jeschke, Verbrennungen: Diagnose, Therapie, Rehabilitation des thermischen Traumas, Springer, Wien New York; 2009; 2, S5- 23
- [Background] Kloth LC. Electrical stimulation for wound healing: a review of evidence from in vitro studies, animal experiments, and clinical trials. Int J Low Extrem Wounds. 2005 Mar;4(1):23-44. doi: 10.1177/1534734605275733. PMID 15860450
- [Background] Mogens, S.; Wirsing, P.; Siemers, F.; Andersen, F. Healing of chronic wound by Wireless Micro Current Stimulation. 2011
- [Background] Sebastian A, Syed F, Perry D, Balamurugan V, Colthurst J, Chaudhry IH, Bayat A. Acceleration of cutaneous healing by electrical stimulation: degenerate electrical waveform down-regulates inflammation, up-regulates angiogenesis and advances remodeling in temporal punch biopsies in a human volunteer study. Wound Repair Regen. 2011 Nov;19(6):693-708. doi: 10.1111/j.1524-475X.2011.00736.x. Epub 2011 Oct 19. PMID 22092840
- [Background] Ud-Din S, Bayat A. Electrical Stimulation and Cutaneous Wound Healing: A Review of Clinical Evidence. Healthcare (Basel). 2014 Oct 27;2(4):445-67. doi: 10.3390/healthcare2040445. PMID 27429287
- [Background] Whelan HT, Smits RL Jr, Buchman EV, Whelan NT, Turner SG, Margolis DA, Cevenini V, Stinson H, Ignatius R, Martin T, Cwiklinski J, Philippi AF, Graf WR, Hodgson B, Gould L, Kane M, Chen G, Caviness J. Effect of NASA light-emitting diode irradiation on wound healing. J Clin Laser Med Surg. 2001 Dec;19(6):305-14. doi: 10.1089/104454701753342758. PMID 11776448
- [Background] Zhao M, Pu J, Forrester JV, McCaig CD. Membrane lipids, EGF receptors, and intracellular signals colocalize and are polarized in epithelial cells moving directionally in a physiological electric field. FASEB J. 2002 Jun;16(8):857-9. doi: 10.1096/fj.01-0811fje. Epub 2002 Apr 10. PMID 11967227
- [Background] Zhao M, Song B, Pu J, Wada T, Reid B, Tai G, Wang F, Guo A, Walczysko P, Gu Y, Sasaki T, Suzuki A, Forrester JV, Bourne HR, Devreotes PN, McCaig CD, Penninger JM. Electrical signals control wound healing through phosphatidylinositol-3-OH kinase-gamma and PTEN. Nature. 2006 Jul 27;442(7101):457-60. doi: 10.1038/nature04925. PMID 16871217